CLINICAL TRIAL: NCT00687427
Title: Return to Work After Hand Injury: The Role of Medical, Demographic and Psychosocial Factors
Brief Title: Return to Work After Hand Injury: the Role of Medical, Demographic and Psycho-Social Factors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Amiram Sagi, Hand Surgery Unit, Soroka University Medical Center
Other Study IDs: sor470708ctil
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Hand Injury
MeSH Terms: conditions — Hand Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (3):
- A: Group A - 25 individuals or more, that start occupational therapy and agree to participate in the research.
  Interventions: Behavioral: Questionnaires and motor/sensitivity testing
- B: Group B- 25 individuals or more, half a year after hand injury that were treated in occupational therapy at the same institute.
  Interventions: Behavioral: Questionnaires and motor/sensitivity testing
- C: Group C - 25 individuals or more, a year after hand injury that were treated in occupational therapy at the same institute
  Interventions: Behavioral: Questionnaires and motor/sensitivity testing

INTERVENTIONS:
Behavioral: Questionnaires and motor/sensitivity testing — Group A:
  1. Full assessment (using the various measures described) will be carried out 0-3 weeks since referral.
  2. Treatment will focus on the patient's needs and in accordance with the physicians requests.
  3. Three months post initial treatment re-assessment will be conducted.
  Groups: A
Behavioral: Questionnaires and motor/sensitivity testing — Group B Researcher will contact by phone previous patients that were treated in the occupational therapy department in the past half year and a year, in order to get their permission to participate (retrospectively) in this research. After getting their consent, a questionnaire concerning their RTW will be posted to the subjects.
  Groups: B
Behavioral: Questionnaires and motor/sensitivity testing — Group C Researcher will contact by phone previous patients that were treated in the occupational therapy department in the past half year and a year, in order to get their permission to participate (retrospectively) in this research. After getting their consent, a questionnaire concerning their RTW will be posted to the subjects.
  Groups: C

SUMMARY:
The purpose of this study is to investigate the extent of return to work (RTW) after traumatic hand injury and to identify factors that are related to RTW.

DETAILED DESCRIPTION:
RTW is one of the main rehabilitation outcomes after injury, the loss of the ability to work may have psychological as well as economic impact on the injured person. Time off work is also a burden to the economic system, associated with loss of work days, sick leave and national insurance payment. Hand injury can cause limitations in function, therefore influence the ability to work. Review of the literature reveals that time off work after hand injury ranges from a few days to a year and more. Factors associated with time off work include medical, socio-economic and psychosocial factors. Only a few studies have been conducted in Israel to investigate rate of RTW after hand injury and factors that affect RTW . The aim of this study is to explore the extent of RTW after traumatic hand injury and to examine the relationship between several factors - medical, demographic and psychosocial and RTW. This, in order to identify prognostic factors that can be treated during rehabilitation. There is no preliminary hypothesis made about the relationships between the factors and RTW. This study is also retrospective and prospective since it examine individuals under-going occupational therapy treatment and individuals who have been treated in the past.

ELIGIBILITY:
Inclusion Criteria:

* The individual worked until he/she was injured
* Traumatic hand injury including: wrist fractures, fingers fractures, tendon injury, nerve injury, Crush injury, finger amputation

Exclusion Criteria:

* Non traumatic hand injury (such as CTS)
* Mallet finger
* Burns
* Injury in several organs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals will be recruited from those referred to occupational therapy department at Soroka Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2008-06; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
RTW vs no RTW | Group A: within 0-3 weeks from referral to occupational therapy treatment and again three months later or at the end of treatment .Group B: half a year after injury. Group C: one year after injury.

SECONDARY OUTCOMES:
Medical, socio-demographic and work environment questionnaires | Group A: within 0-3 weeks from referral to occupational therapy treatment and again three months later or at the end of treatment .Group B: half a year after injury. Group C: one year after injury.
psychosocial questionnaires including: Post Traumatic Stress Disorder questionnaire, McGill Pain Questionnaire, pain belief and self-efficacy questionnaires. | Group A: within 0-3 weeks from referral to occupational therapy treatment and again three months later or at the end of treatment .Group B: half a year after injury. Group C: one year after injury.
Motor and sensitivity testing : hand grip and pinch strength measurements, Purdue Pegboard Test, Semmes-Weinstein Pressure Monofilaments, upper extremity rang of motion, Pain Visual Analogue Scale. | within 0-3 weeks from referral to occupational therapy treatment and again three months later or at the end of treatment .
Disabilities of Arm Shoulder and Hand questionnaire | Group A: within 0-3 weeks from referral to occupational therapy treatment and again three months later or at the end of treatment .Group B: half a year after injury. Group C: one year after injury.

CONTACTS AND LOCATIONS:
Overall Officials: Amiram Sagi, Professor, Principal Investigator — Hand Surgery Unit, Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Occupational Therapy Department, Beersheba, Israel

REFERENCES:
- [Background] Bear - Lehman, J. (1983). Factors Affecting Return to Work After Hand Injury. American Journal of Occupational Therapy, 37 (3), 189 - 194. Chan, J., & Spencer, J. (2004). Adaptation to Hand Injury: An Evolving Experience. American Journal of Occupational Therapy, 58 (2), 128 - 139. Chan, J., & Spencer, J. (2005). Contrasting Perspectives on Pain following Hand Injury. Journal of Hand Therapy, Oct-Dec 18 (4),429 - 436. Chen, C.Y., Strecker Neufeld, P., Feely, C.H., & Skinner C.S. (1999). Factors Influencing Compliance With Home Exericise Programs Among Patients With Upper Extremity Impairment. American Journal of Occupational Therapy, 53 (2), 171 - 180. Deem, R. (1988). Work, Unemployment and Leisure. London: Routledge. DeGood, D.E., & Shutty, M.S. (1992). Assessment of Pain Beleifs, Coping, ans Self Efficancy. In D.C. Turk ,& R. Melzack (Eds), Hand Book of Pain Assessment, pp. 214 - 230. New York: The Guilford . Flood, A.B., Loernce, D.P., Ding, J., McPherson, K., & Black, N.A. (1993). The Role of Expectations in Patient's Reports of Post-Operative Outcomes and Improvement Following Therapy. Medical Care, 31 (11), 1043 - 1056. Franche R.L. & Krause N. (2002) Readiness for Return to Work Following Injury or Illness: Conceptualizing the Interpersonal Impact of Health Care, Workplace, and Insurance Factors. Journal of Occupational Rehabilitation,12 (4), 233 - 256. Gage, M. N., & Polatajko, H. (1994). Enhanching occupational performance through an understanding of percieved self-efficacy. American Journal of Occupational Therapy, 48, 452 - 461. Grunert, B.K., Matloub, H.S., Sanger, J.R., & Yousif, N.J. (1990). Treatment of Posttraumatic Stress disorder after work-related hand trauma. The Journal of Hand Surgery, 15A (3), 511 - 515. Jensen, P.J., Turner, J.A., Romano, J.M., & Lawler, B.K. (1994). Relationship of pain-specific beliefs to chronic pain adjustment. Pain , 57, 301 - 309. Johns, A.M. (1981). Time off work after hand injury. Injury ,Mar 12 (5), 417 - 424. Kasdan, M.L., & June, L.A. (1993). Returning to Work after Unilateral Hand Fracture. Journal of Occupational Medicine, 35(2), 132 - 136. Kelvin, P. & Jarret, J.E. (1985). Unemployment its social psychological effects. Cambridge University Press. Kilhofner, G. (2002). A Model of Human Occupation: Theory and Application (3 ed). Baltimore: Lippincott Williams & Wilkins. Krause, N., Frank, J.W., Dasinger, L.K., Sullivan. T.J., & Sinclair, S.J. (2001). Determinants of Duration of Disability and Return to Work after Work-Related Injury and Illness: Challenges for Future Research. American Journal of Industrial Medicine, 40, 464 - 484. Lai, C.H. (2004). Motivation in Hand-injured Patient with and without Work-related Injury. Journal of Hand Therapy, Jan-Mar 17 (1), 6 - 17. Melamed, S., Grosswasser, Z., & Stern, M.J. (1992). Acceptance of disability, work involvemnt and subjective rehabilitation status of traumatic brain injured (TBI) patients. Brain Injury, 6, 233 - 243. Mink Van Der Molen, A.B., Groothoff, J.W., Visser, J.P., Robinson, P.H., & Eisma, W.H. (1999). Time off Work due to Scaphoid Fracture and other Carpal Injuries in the Netherlands in the period 1990 to 1993. Journal of Hand Surgery (British and European Volume), 24b (2), 193-198. Pransky, G., Gatchel, R., Linton, S.J., & Loisel, P. (2005). Improving Return to Work Research. Journal of Occupational Rehabilitation, 15(4), 453 - 457. Rainwater, L. (1974). Work, Well-Being, and Family Life. In J. O'Toole (Ed), Work and the Quality of life, pp361-370. Cambridge Mass: Mit Press Rosberg, H.E., Steen-Carlsson, K., & Dahlin, L.B. (2005). Prospective study of patients with injuries to the hand and forearm: cost, function and genral health. Scandinavian journal of plastic and reconstructive surgery and hand surgey, 39 (6), 360-369. Rusch, M.D., Dzwierzynski, W.W., Sanger, J.R., Pruit, N.T., Siewert, A.D. (2003). Return to Work Outcomes after Work-Related Hand Trauma: The Role of Causal Attributions. The Journal of Hand Surgery, 28A, No. 4, 673 - 677. Schultz-Johnson, K. (1987). Assessment of Upper Extremity-injured persons' return to work potentail. Journal of Hand Surjery, 12A (5), 950 - 957. Skov, O., Jeune. B., Lauritsen J.M., & Barfred, T. (1999). Time off Work After Occupational Hand Injuries. Journal of Hand Surgery (British and European Volume), 24B (2): 187 - 189. Waylett-Rendall, J., & Niemeyer, L.O. (2004). Exploratory Analysis to Identify Factors Impacting Return-to-Work Outcomes in Cases of Cumulative Trauma Disorder. Journal of Hand Therapy, Jan-Mar, 17(1), 50 - 57.